CLINICAL TRIAL: NCT00567008
Title: A Double-Blind Placebo-Controlled Pilot Trial of Varenicline (Chantix) for the Treatment of Cocaine Dependence
Brief Title: Chantix for Treating Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jennifer Plebani, Jennifer Plebani, PhD, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 806565; P60DA005186 (NIH); NIDA P60DA0005186
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Results first posted 2013-11-07 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-10

CONDITIONS: Cocaine Dependence
Keywords: cocaine; crack cocaine; cocaine-related disorders; substance-related disorders; alpha4beta2 nicotinic acetylcholine receptor
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Varenicline (Chantix)
  Interventions: Drug: varenicline
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varenicline — 1.0 mg BID for 8 weeks
  Other Names: Chantix
  Arms: 1
Drug: placebo — placebo BID for 8 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether varenicline (Chantix), is effective for the treatment of cocaine dependence.

DETAILED DESCRIPTION:
The purpose of study is to determine if Varenicline (Chantix™) promotes cocaine abstinence in cocaine dependent individuals. Varenicline (Chantix™) (2.0 mg/day) or placebo will be administered in a 9-week double-blind trial to patients meeting diagnostic criteria for cocaine dependence.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 to 65 years old.
* Meets DSM-IV criteria for Cocaine Dependence, as determined by the Structured Clinical Interview for DSM-IV (SCID).
* Live within a commutable distance of the Treatment Research Center (TRC) at the Penn/VA Center for Studies of Addiction, University of Pennsylvania. We define this to be a distance within the service area of Septa, within an hour drive, or a distance that both the patient and Principal Investigator (PI) find acceptable.
* Understands and signs the informed consent.

Exclusion Criteria:

* Current DSM-IV diagnosis of any psychoactive substance dependence other than cocaine or nicotine dependence, as determined by the SCID.
* Concomitant treatment with psychotropic medications.
* Current or prior gambling problems. This will be assessed by the patient's self-report.
* Patients mandated to treatment based upon a legal decision or as a condition of employment. This will be assessed by the patient's self-report.
* Current severe psychiatric symptoms, e.g., psychosis, dementia, suicidal or homicidal ideation, mania or depression requiring antidepressant therapy in the opinion of the Principal Investigator (PI)
* Use of any investigational medication within the past 30 days.
* History of significant heart disease (an arrhythmia which required medication, Wolff-Parkinson -White Syndrome, angina pectoris, documented history of myocardial infarction, heart failure).
* History of chest pain associated with cocaine use that has prompted a visit to a physician.
* Current use of naltrexone, disulfiram, modafinil, stimulants, reserpine, verapamil, theophylline, trimethoprim, cimetidine, haloperidol, benzodiazepines or anticonvulsants.
* Known hypersensitivity to varenicline.
* Patients with known AIDS or other serious illnesses that may require hospitalization during the study.
* Female subjects who are pregnant or lactating, or female subjects of child-bearing potential who are not using acceptable methods of birth control.

Acceptable methods of birth control include:

* barrier (diaphragm or condom) with spermicide
* intrauterine progesterone contraceptive system
* levonorgestrel implant
* medroxyprogesterone acetate contraceptive injection
* oral contraceptives.
* tubal ligation.
* Patients with impaired renal function as indicated by corrected creatinine clearance below 80 ml/min/70 kg as determined by the modified Cockcroft equation (CDC, 1986).
* Clinical laboratory tests (CBC, blood chemistries, urinalysis) outside normal limits that are clinically unacceptable to the Principal Investigator. EKG 1st degree heart block, sinus tachycardia, left axis deviation, and nonspecific ST or T wave changes are allowed; liver function tests [LFTs] <5 x ULN are acceptable).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer G Plebani, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-seven treatment-seeking participants from the greater metropolitan Philadelphia area were randomized to participate in this trial.
Groups:
- Varenicline 2mg/Day: Varenicline (Chantix)
- Placebo: Placebo
Period: Overall Study
Arm/Group | Varenicline 2mg/Day | Placebo
Started | 18 | 19
Completed | 17 | 18
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Varenicline: Varenicline (Chantix)
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 13 | 14 | 27
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Abstinence From Cocaine as Indicated by Qualitative Urinalysis for Benzoylecgonine.
Description: Number of Participants that Tested Negative for Benzoylecgonine in Qualitative Urinalysis Assessment.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 18 | 19
participants | 2 [lower limit 0.91] | 1

ADVERSE EVENTS:
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 15/17 | 17/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=17) | Placebo (N=18)
Headache (General disorders) | 3 (4) | 5 (7)
Body aches/paines (General disorders) | 3 (5) | 8 (12)
Cold (Gastrointestinal disorders) | 4 (4) | 0 (0)
Drowsiness (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 5 (5)
Cough (General disorders) | 2 (3) | 1 (1)
Nighmare (General disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 3 (3)
Insomnia (General disorders) | 2 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was a small preliminary trial, and thus was underpowered for anything less than large effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No